CLINICAL TRIAL: NCT05145959
Title: Meibomian Gland Probing in the Sub-Acute Phase of Patients With Stevens-Johnson Syndrome/Toxic Epidermal Necrolysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Hajirah N. Saeed, M.D., Principal Investigator, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P000608
Record Dates: First submitted 2021-10-21; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Stevens-Johnson Syndrome; Toxic Epidermal Necrolyses; Ocular Surface Disease; Meibomitis; Meibomian Gland Dysfunction; Dry Eye
Keywords: Stevens-Johnson Syndrome
MeSH Terms: conditions — Stevens-Johnson Syndrome; Meibomitis; Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Maskin Probe — The eyelids are examined using meibography to evaluate which eyelids are more severe (right or left). A drop of proparacaine 0.5% solution is added and a bandage contact lens is placed. To avoid patient discomfort, anesthetic ointment is instilled using a sterile cotton-tipped applicator. In some cases, 4% lidocaine can be directly applied to the lid margin. The Maskin probe will be passed through the gland orifice perpendicular to the lid margin. After first using a 1-mm probe, a 2- or 4-mm probes may be used in cases of persistent resistance. The BCL is removed and the eyes are rinsed with sterile preservative-free saline. The patient is given preservative-free artificial tears to use every hour. A brief slit lamp exam will performed in order to ensure that there is no unanticipated damage to the lid or cornea. The probing device will be properly disposed of in the sharps containers.

SUMMARY:
The investigators' aim is to study the effects of mechanical expression of meibomian glands on eyelid disease, ocular surface health in the subacute phase of SJS/TEN.

The primary outcome is to use meibomian gland imaging to assess the health and caliber of the meibomian glands of both lower eyelids, between the treated and non-treated eyes before and after the intervention. Monitoring of outcomes will be measured by comparing the results of meibography at the initial visit and at the 6-month follow-up.

The secondary outcome assessed will be patient symptoms. The Ocular Surface Disease Index survey will be administered before each treatment and patients will be asked to differentiate their symptoms between the two eyes, both before and after the intervention.

The investigators hypothesize that mechanical expression of meibomian glands within the first 6 months of SJS/TEN onset will significantly improve ocular surface disease and symptoms in those patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SJS/TEN presenting to the Massachusetts Eye and Ear Infirmary (MEEI) ophthalmology clinic or who were seen by the ophthalmology team acutely at the Massachusetts General Hospital (MGH).
* Patients must be in the Sub-acute phase of ocular SJS (within 6 months)
* Patients must have evidence of Meibomitis
* Patients must be adults (18 years of age or older)

Exclusion Criteria:

* Patients with unconfirmed diagnosis of SJS vs. Erythema multiforme (or other condition).
* Patients beyond the sub-acute phase of SJS
* Patients without evidence of Meibomitis (See above criteria)
* Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Meibomian gland imaging (Meibography) - Qualitative description | 6 months
  To assess the appearance of the meibomian glands of both lower eyelids, before and after the intervention.

SECONDARY OUTCOMES:
Ocular Surface Disease Index survey | 6 months
  The Ocular Surface Disease Index survey will be administered before each treatment and patients will be asked to differentiate their symptoms between the two eyes, both before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts Eye and Ear Hospital, Boston, Massachusetts, United States